CLINICAL TRIAL: NCT07285083
Title: Comparison of Pain Relief by Bupivacaine With Dexmedetomidine and Bupivacaine Alone in Transversus Abdominis Plane Block for Postoperative Analgesia in Patients Undergoing Abdominal Surgeries.
Brief Title: Bupivacaine With or Without Dexmedetomidine for Postoperative Pain Relief in Abdominal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheikh Zayed Medical College (Other Government)
Responsible Party: Principal Investigator, Rameesha Musharaf, POST GRADUATE RESIDENT (ANESTHESIA), Sheikh Zayed Medical College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 696/IRB/SZMC/SZH
Record Dates: First submitted 2025-11-20; First posted 2025-12-16 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-11

CONDITIONS: Pain, Postoperative
Keywords: Transversus abdominis plane (TAP) block
MeSH Terms: conditions — Pain, Postoperative; Bites and Stings | interventions — Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial (RCT) where patients are assigned to one of two groups. Group A will receive bupivacaine with dexmedetomidine, and Group B will receive only bupivacaine via a transversus abdominis plane (TAP) block. The primary outcome is pain relief measured by the Visual Analogue Scale (VAS).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: This study will use a double-blind design, where both the participants and care providers (including anesthesiologists) are unaware of the treatment allocation. The outcomes assessors are also blinded to ensure unbiased pain assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine + Dexmedetomidine (TAP Block) (Experimental): Participants in this arm will receive a combination of 20 ml of 0.25% bupivacaine and 1 mcg/kg dexmedetomidine administered via an ultrasound-guided transversus abdominis plane (TAP) block for postoperative pain management following abdominal surgery
  Interventions: Drug: Bupivacaine (TAP Block)
- Bupivacaine Only (TAP Block) (Active Comparator): Participants in this arm will receive 20 ml of 0.25% bupivacaine administered via an ultrasound-guided transversus abdominis plane (TAP) block for postoperative pain management following abdominal surgery
  Interventions: Drug: Bupivacaine with Dexmedetomidine (TAP Block)

INTERVENTIONS:
Drug: Bupivacaine with Dexmedetomidine (TAP Block) — A combination of 0.25% bupivacaine and 1 mcg/kg dexmedetomidine administered bilaterally via ultrasound-guided transversus abdominis plane (TAP) block to provide postoperative analgesia for abdominal surgery
  Arms: Bupivacaine Only (TAP Block)
Drug: Bupivacaine (TAP Block) — 10 ml of 0.25% bupivacaine administered bilaterally via ultrasound-guided transversus abdominis plane (TAP) block to provide postoperative analgesia for abdominal surgery
  Arms: Bupivacaine + Dexmedetomidine (TAP Block)

SUMMARY:
This study investigates the effectiveness of adding dexmedetomidine to bupivacaine for postoperative analgesia in patients undergoing abdominal surgeries. The research compares pain relief in two groups: one receiving a combination of bupivacaine and dexmedetomidine via a transversus abdominis plane (TAP) block, and the other receiving bupivacaine alone. The study aims to evaluate whether dexmedetomidine enhances pain relief, reduces the need for additional pain medication, and impacts sedation and side effects such as hypotension, bradycardia, and nausea. Conducted at Sheikh Zayed Medical College in Rahim Yar Khan, Pakistan, the trial will involve 80 participants and will measure pain using the Visual Analogue Scale (VAS), along with monitoring other vital parameters and complications over 12 hours post-surgery. The primary objective is to determine if the addition of dexmedetomidine provides superior pain control without significantly increasing side effects.

DETAILED DESCRIPTION:
This randomized controlled trial will assess the comparative effectiveness of bupivacaine with and without dexmedetomidine in managing postoperative pain following abdominal surgeries. The study will be conducted at Sheikh Zayed Medical College and Hospital, Rahim Yar Khan, Pakistan. A total of 80 patients, aged 21-45 years, undergoing elective abdominal surgeries will be included. These participants will be randomly divided into two groups: Group A will receive a combination of bupivacaine and dexmedetomidine, and Group B will receive only bupivacaine.

The primary outcome is pain relief, assessed using the Visual Analogue Scale (VAS) at multiple time points. Secondary outcomes include the Ramsay Sedation Score, heart rate, mean arterial pressure, and the occurrence of side effects such as hypotension, bradycardia, and nausea. Rescue analgesia will be provided if the VAS score exceeds 4. Both groups will receive ultrasound-guided TAP blocks at the end of their surgeries.

The study aims to evaluate whether the addition of dexmedetomidine improves the duration of analgesia and reduces the need for additional analgesics without exacerbating side effects. The null hypothesis is that there will be no significant difference in pain relief between the two groups, while the alternative hypothesis is that dexmedetomidine will provide superior analgesia.

Statistical analysis will be performed using SPSS v23, with a significance level set at p < 0.05. Data will be analyzed for both quantitative outcomes (e.g., pain scores, heart rate, blood pressure) and qualitative outcomes (e.g., side effects). Stratification by age, gender, and comorbidities will control for potential confounding variables.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 21 to 45 years.
2. Undergoing elective abdominal surgery (exploratory laparotomy, ileostomy reversal, laparoscopic/open cholecystectomy, mesh repair of paraumbilical hernias).
3. The patient must be capable of providing informed consent.

Exclusion Criteria:

1. Pregnancy.
2. Severe allergies to local anesthetics.
3. Pre-existing chronic pain conditions.
4. Participation in another clinical trial within the past 30 days.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Relief (Visual Analogue Scale - VAS) | Time Frame: 1-12 hours post-surgery.
  The primary outcome is postoperative pain level, measured using the Visual Analogue Scale (VAS), a 10-point scale ranging from 0 to 10, where 0 = no pain and 10 = worst pain imaginable. Higher scores indicate worse pain. Pain scores will be recorded at 1, 3, 6, 9, and 12 hours post-surgery.

SECONDARY OUTCOMES:
Sedation Level (Ramsay Sedation Scale) | Time Frame: Up to 12 hours post-surgery.
  Sedation level will be assessed using the Ramsay Sedation Scale, which ranges from 1 to 6, where 1 = anxious/agitated and 6 = no response to stimuli. Higher scores indicate deeper sedation. Measurements will be recorded at 15 minutes, 30 minutes, and 1, 3, 6, 9, and 12 hours post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Saira Sadaf, FCPS ANESTHESIA, Study Chair — Shaheed Ziaur Rahman Medical College
Locations (1):
- Sheikh Zayed Medical College, Rahim Yar Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
The study will not share individual participant data (IPD) due to the sensitive nature of the data and the lack of a formal data-sharing agreement. The study aims to protect patient confidentiality and privacy. As such, the data will only be used for the purpose of this trial and will not be made available to external researchers.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/83/NCT07285083/Prot_SAP_000.pdf